CLINICAL TRIAL: NCT05877820
Title: A Prospective, Single Arm Clinical Study to Evaluate Efficacy and Safety of Lenvatinib Combined With Tislelizumab in the First Line Treatment of Patients With Locally Advanced or Metastastic Fumarate Hydratase Deficient Renal Cell Carcinoma
Brief Title: A Study to Evaluate Efficacy and Safety of Lenvatinib Combined With Tislelizumab in Patients With FHRCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LENTIS
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Fumarate Hydratase Deficient Renal Cell Carcinoma
Keywords: PD-1 checkpoint inhibitor; FHRCC
MeSH Terms: interventions — tislelizumab; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab+Lenvatinib combination therapy (Experimental): Participants receive tislelizumab 200 mg intravenously every 3 weeks PLUS lenvatinib 20mg orally once daily.
  Interventions: Biological: Tislelizumab; Drug: Lenvatinib

INTERVENTIONS:
Biological: Tislelizumab — Intravenous infusion
Drug: Lenvatinib — Oral tablet

SUMMARY:
FHRCC is a rare kind of renal cell carcinoma with a morbidity of 1/2000000 per year.Although several combination therapies demonstrated possible efficacy in this population. No standard treatment has been approved. The purpose of this study is to evaluate the efficacy and safety of Lenvatinib in combination with tislelizumab in the first line treatment of patients with locally advanced/metastatic FHRCC.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand and voluntarily sign the informed consent form and agree to receive treatment, examination and follow-up as required by the study protocol;
2. Age ≥ 18, < 80 years, male or female;
3. ECOG score ≤2;
4. unresectable or recurrent metastatic FH-deficient renal cell carcinoma not previously treated with systemic antitumor therapy, as confirmed by histology. Prior cytokine therapy is allowed;
5. At least 1 measurable tumor lesion according to RECIST 1.1 criteria. The lesion that has received prior radiotherapy and progressed again is allowed as a target lesion;
6. agree to provide blood and urine samples and previous archived or fresh tumor tissue samples.
7. Demonstrates adequate organ function.
8. Female subjects of childbearing potential must have a negative serum pregnancy test result within 7 days prior to the first dose. participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 180 days after the last dose of study drug.

Exclusion Criteria:

1. Prior treatment with agents targeting VEGF, VEGFR, or mTOR, including but not limited to sunitinib, axitinib, pazopanib, sorafenib, cabozantinib, lenvatinib, bevacizumab, anlotinib, or everolimus;
2. Prior treatment with anti-PD-1, PD-L1 or CTLA-4 antibodies;
3. Participants who are using other investigational agents or who had received investigational drugs <=4 weeks prior to study treatment start;
4. Received major surgery or is recovering from surgery (as judged by the investigator) within 4 weeks;
5. Received Chinese herbal or proprietary Chinese medicine preparation with an antitumor indication within 2 weeks;
6. Requirement of adrenocorticosteroids (>10 mg prednisone or equivalent daily) or other immunosuppressive systemic therapy within 2 week; inhalation of >10 mg prednisone or equivalent daily, but without active autoimmune disease may participate in this study;
7. History of organ transplantation or conditions requiring long-term adrenocorticosteroid or immunosuppressive therapy
8. Hypothyroidism, adrenal or pituitary gland function that can be controlled with hormone replacement therapy, type I diabetes mellitus, psoriasis or vitiligo that do not require systemic therapy may be enrolled in the study;
9. Didn't recover from prior antineoplastic therapy, grade 0 to 1 as defined by NCI-CTCAE 5.0 (except alopecia), or levels specified in the inclusion/exclusion criteria. Irreversible toxicity that is not expected to be exacerbated by the study drug can be enrolled;
10. The presence of other malignancies that have progressed or require treatment within 5 years (excluding basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer or cured carcinoma in situ, such as carcinoma in situ of the breast, prostate cancer: subjects with limited low-risk prostate cancer (≤ T2a, Gleason score ≤ 6, PSA < 10ng/ml) who have received radical treatment and no PSA biochemical (those with recurrence may participate in this study);
11. History of active central nervous system (CNS) metastases or baseline phase imaging showing CNS metastases within 30 days prior to the first dose. Subjects with prior surgical or radiation treatment for brain or meningeal metastases who have maintained clinical stability for ≥ 3 months by screening and have discontinued systemic hormone therapy (dose > 10 mg/day of prednisone or other equivalent hormone) for > 4 weeks may be enrolled. Subjects may be enrolled in this study if the subject's CNS metastases can be treated to meet the requirements of the enrollment criteria and if the subject's CNS symptoms have returned to ≤ grade 1 for at least 2 weeks prior to enrollment (except for residual signs or symptoms related to CNS treatment);
12. Poorly controlled hypertension: SBP ≥ 150 mmHg and/or DBP ≥ 90 mmHg;
13. Any one or more of the following cardiovascular disease states within the last 6 months: myocardial infarction; unstable angina; endoluminal angioplasty or coronary stenting; coronary/peripheral artery bypass graft; NYHA cardiac function class 3-4; congestive heart failure; cerebrovascular accident including transient ischemic attack;
14. Heart rate corrected QT interval (QTc) ≥ 480 ms;
15. History of active bleeding or other severe bleeding within 1 month;
16. Deep vein thrombosis or pulmonary embolism within 6 months;
17. Arterial embolism within the last 12 months;
18. Clinically significant gastrointestinal abnormalities, including: malabsorption, total gastrectomy, or any condition that may interfere with the absorption of oral medications; active ulcers treated within 6 months; active gastrointestinal bleeding (vomiting blood, blood in stool, or black stool) within 3 months by endoscopy; metastatic lesions in the gastrointestinal tract suspected of bleeding, inflammatory bowel disease, ulcerative colitis Gastrointestinal perforation or other gastrointestinal disorders that increase the risk of perforation;
19. The presence of (non-infectious) pneumonia/interstitial lung disease requiring adrenocorticosteroid therapy, either previously or currently
20. Presence of active infection requiring systemic therapy, presence of human immunodeficiency virus (HIV) infection (known HIV antibody positivity), presence of active HBV infection (HBsAg positive, or HBcAb positive but HBsAg negative, additional DNA quantification is required and results that do not exceed the upper limit of normal laboratory values can be enrolled), presence of active HCV infection (previous HCV infected patients with negative HCV RNA test results during the screening period can be enrolled);
21. Live virus vaccinations within the last 1 month, including but not limited to mumps, rubella, measles, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccines, excluding inactivated virus vaccines;
22. A history of severe drug allergy, including but not limited to antibody drugs and small molecule targeted drugs;
23. Known psychiatric illness or history of substance abuse;
24. Presence of unhealed wounds;
25. The presence of any medical history or current evidence of disease, treatment or laboratory abnormality that, in the investigator's judgment, could confound the results of the trial, interfere with the subject's participation in the full trial, or is not in the subject's best interest to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 24 months
  ORR was determined per RECIST 1.1 and was defined as the percentage of participants in the analysis population who had a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 24 months
  PFS was defined as the time from enrollment to the first documented progressive disease (PD) or death due to any cause, whichever occurred first.
Overall Survival (OS) | Up to approximately 24 months
  OS was defined as the time from enrollment to death due to any cause.
Disease Control Rate (DCR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 24 months
  DCR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions), Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters), or Stable Disease (SD) per RECIST 1.1 for ≥6 months.
Duration of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 24 months
  DOR was defined as the time from first documented evidence of a Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1 until progressive disease (PD) or death due to any cause, whichever occurred first.
Overall Survival (OS) Rate at Month 12 in All Participants | Month 12
  The OS rate was determined for all participants at Month 12 and was defined as the time from enrollment to death due to any cause.
Overall Survival (OS) Rate at Month 24 in All Participants | Month 24
  The OS rate was determined for all participants at Month 24 and was defined as the time from enrollment to death due to any cause.
Number of Participants Who Experienced an Adverse Event (AE) | Up to approximately 24 months
  An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of Shanghai Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD